CLINICAL TRIAL: NCT02999529
Title: Improving Patient Understanding of Key Terms Used to Describe Chemotherapy and Its Side Effects
Brief Title: Health Literacy Multi-media Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rebecca D. Pentz, PhD, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00085515
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Cancer
Keywords: Chemotherapy; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Education Group (Experimental): Participants offered a consent for chemotherapy treatment will watch an educational video.
  Interventions: Other: Educational Video

INTERVENTIONS:
Other: Educational Video — Participants will be asked if they know the meaning of six words related to cancer treatment. Following the interview, participants will watch a video explaining the meaning of the six words. After viewing the video, participants will be re-interviewed about the meaning of the six words.

SUMMARY:
Cancer patients are presented with a lot of information about their diagnosis and different treatment options, which can be confusing. The purpose of this study is to see if a simple video explanation of six words used to describe cancer treatment improves patient understanding of these words.

DETAILED DESCRIPTION:
Cancer patients are presented with a lot of information about their diagnosis and different treatment options, which can be confusing. The purpose of this study is to see if a simple video explanation of six words used to describe cancer treatment improves patient understanding of these words.

Participants will be interviewed and asked the meaning of six words related to cancer treatment. Following the interview, participants will be shown a video about the meaning of the words. After viewing the video, participants will be re-interviewed to test how effective the video was at explaining the six words.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Grady Memorial Hospital who is offered a consent to receive chemotherapy

Exclusion Criteria:

* Profession as a physician or nurse
* Non English speaking

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Number of Correct Responses | Post Intervention (Up to ten minutes)
  The number of correct responses to the meaning of the six cancer treatment words will be collected after watching the educational video.
Number of Incorrect Responses | Post Intervention (Up to ten minutes)
  The number of incorrect responses to the meaning of the six cancer treatment words will be collected after watching the educational video.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Pentz, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States